CLINICAL TRIAL: NCT00965666
Title: Etanercept (Enbrel) in Children With Fanconi Anemia and Early Bone Marrow Failure: A Pilot Study
Brief Title: Pilot Study of Etanercept (Enbrel) in Children With Fanconi Anemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-07-24
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2012-03

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia; Hemic and Lymphatic Diseases; Anti-Rheumatic Agents; Anemia, Hypoplastic, Congenital; DNA Repair-Deficiency Disorders; Congenital, Hereditary, and; Neonatal Diseases and Abnormalities
MeSH Terms: conditions — Fanconi Anemia; Hemic and Lymphatic Diseases; Anemia, Hypoplastic, Congenital; DNA Repair-Deficiency Disorders; Congenital, Hereditary, and Neonatal Diseases and Abnormalities | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — All qualified subjects receive 24 weekly subcutaneous injections of Etanercept.
  Other Names: Enbrel

SUMMARY:
The purpose of this research study is to evaluate the safety of the drug Etanercept (Enbrel) and to determine if this drug can help in the treatment of early bone marrow failure in patients with Fanconi anemia.

DETAILED DESCRIPTION:
Patients with FA are treated with blood products (transfusions), injections to stimulate white blood cell production, and/or androgen therapy once they reach advanced stages of bone marrow failure. Although these therapies lead to temporary improvement in the blood counts, they are associated with potential serious side effects. Currently, the only known potential cure for bone marrow failure in Fanconi Anemia is a stem cell transplant, which is usually done at the late stages of bone marrow failure and is again associated with significant toxicity.

Studies show that patients with FA are very sensitive to and produce unusually high levels of a protein called tumor necrosis factor alpha (TNF-α) that causes bone marrow cells to die. We will study whether a drug called Etanercept that reduces levels of TNF-α will delay or prevent the progressive bone marrow failure associated with FA. Etanercept has been successfully used in children with arthritis.

Primary Objectives:

1. To assess toxicity of Etanercept (Enbrel) in children with Fanconi Anemia (FA) and early marrow failure.
2. To assess efficacy of Etanercept (Enbrel) in improving hematopoiesis (i.e. peripheral counts) in patients with FA.

Secondary Objectives:

1) Correlation of biological studies to measure the impact of Etanercept (Enbrel) on Tumor Necrosis Factor - α (TNF-α) production.

Fanconi anemia (FA) is an autosomal recessive disease characterized by progressive bone marrow failure, variable congenital abnormalities and a predisposition to malignancy, particularly acute myeloid leukemia (AML) 1. Cells from FA patients exhibit hypersensitivity to alkylating agents such as mitomycin C and diepoxybutane (DEB). Currently, FA is diagnosed by testing for chromosome breakage after lymphocyte stimulation and exposure to mitomycin C (MMC) or diepoxybutane (DEB) 2. Chromosome fragility, defined by an increased percentage of chromosome breaks, is diagnostic for FA3. Although it is the most common form of constitutional aplastic anemia it is very uncommon and the true incidence of FA is not known. A total of 754 patients from North America with the DEB confirmed diagnoses of FA were registered into the International Fanconi Anemia registry (IFAR) by 2001. The major cause of morbidity and mortality for children with FA is bone marrow failure that occurs in the majority of children in the first and second decades of life. Attempts to culture bone marrow progenitors in vitro from FA patients demonstrate decreased numbers of myeloid and erythroid colonies, which is consistent with clinical bone marrow failure.

Current treatment for FA relies upon hematological support in the form of transfusions once advanced marrow failure occurs. Patients with FA do not respond to anti-thymocyte globulin or cyclosporine (typical treatments for acquired aplastic anemia), but 50% improve with androgen preparations, with a median prolongation of life of 2 years in responders (from 16 years to 18 years of age at death) although relapses are inevitable. Androgen therapy causes significant liver toxicity, virilization and risk of hepatic adenoma or carcinoma. Patients who do not respond to these modalities are treated with stem cell transplantation, with its associated toxicities from the transplant conditioning regimens, graft-versus-host disease and increased risk of post transplant malignancy compared to patients without FA. Five-year survival after a matched sibling transplant is approximately 65%. After an unrelated donor transplant, five-year survival is about 30%. The natural history of this disease is one of eventual death by age 10 to 20 years from progressive marrow failure or from conversion to AML (in approximately 10% of patients). Thus there is clearly a need for an effective and early therapy with better toxicity profile.

Studies in both animals and human subjects indicate that high levels of systemic TNF-α and increased sensitivity of hematopoietic progenitors to TNF-α plays a key role in pathogenesis of bone marrow failure in patients with FA. This suggests a possible benefit in supporting hematopoiesis with anti-TNF-α receptor Fc fusion protein (Etanercept; Enbrel) in children with FA. This study proposes to treat patients with FA and early marrow failure with Etanercept (Enbrel), a medication used to treat rheumatoid arthritis. The results of the proposed project will use important preclinical data (see below) to support the development of a novel therapeutic approach for treatment of marrow failure in FA. Etanercept (Enbrel) will prevent the progressive marrow failure and associated complications without the need for transplant and if found to be effective, this treatment can be included in standard clinical care of FA patients, potentially for many years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of FA proven by a DEB test conducted in the cytogenetics lab of Dr. Arleen Auerbach, Rockefeller University Hospital.
2. Patients must have evidence of early marrow failure i.e. reduction in at least one cell line on two separate occasions at least one month apart e.g. platelet count of < 100,000 per cubic millimeter, hemoglobin < 9 gm/dl and/or absolute neutrophil count (ANC) of < 1000
3. Negative pregnancy test (conducted via serum β-HCG screen) - done before the first dose of study drug in all women (except those surgically sterile, at least 5 years postmenopausal, or under the age of 10 years)
4. Sexually active patients of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study
5. Patients or designees must have the ability to self-inject investigational product or have a care giver at home who can administer subcutaneous injections
6. Patients or designees must be able and willing to give written informed consent and comply with the requirements of the study protocol and must authorize release and use of protected health information
7. Patients must have a negative TB skin test at entry into the study

Exclusion Criteria:

1. Patients < 4 yrs of age
2. Patients with advanced marrow failure i.e. transfusion dependent, will not be eligible as we anticipate that stem cell depletion will already be advanced at this stage.
3. Patients currently enrolled in another investigational device or drug trial(s) (defined as a drug not approved by the FDA), or who have received other investigational agent(s) within 28 days of baseline visit with the exception of CCHMC IRB protocol # 03-9-11, "Thyroid Hormone in Children with Fanconi Anemia"
4. Patients on androgen therapy
5. Patients who have received immunosuppressive agents within the last 3 months prior to enrollment
6. Patients who have any grade 3 or 4 adverse event or laboratory toxicity other than in Blood or Bone Marrow (as per the NCI CTC criteria) at the time of the screening visit or at any time during the study, that in the opinion of the Investigator would preclude participation in the study
7. Patients with active infections within 4 weeks before the screening/baseline visit
8. Patients with untreated Lyme disease
9. Patients with a recent or past history of fungal infection
10. Patients who have history of TB or TB exposure, chronic hepatitis B or hepatitis C, SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy
11. Patients with known hypersensitivity to Etanercept (Enbrel) or any of its components or who are known to have antibodies to Etanercept (Enbrel).
12. Patients who have received hematopoietic growth factor for greater than 3 consecutive days in the 6 months before study enrollment (i.e., erythropoietin, filgrastim, neupogen, sargramostin) for clinical purposes to improve bone marrow function. Patients receiving hematopoietic growth factor for stem cell mobilization and collection only are not excluded from this study.
13. Patients with an available matched sibling donor and clinically indicated need for bone marrow transplant
14. Patients with renal failure requiring dialysis
15. Patients with a total bilirubin >3 mg/dl and/or SGPT >200 at time of enrollment
16. Patients who are pregnant or breastfeeding or are a female at risk of pregnancy and are unable to practice safe sex during the length of the study
17. Patients who are HIV positive
18. Patients with severe co-morbidities (diabetes mellitus requiring insulin, CHF of any severity, MI, CVA or TIA within 3 months of screening visit, unstable angina pectoris, uncontrolled hypertension, oxygen-dependent severe pulmonary disease, history of cancer within 5 years (other than resected cutaneous basal or squamous cell carcinoma or in situ cervical cancer)
19. Patients who have any mycobacterial disease or known history of any other immuno-suppressing disease
20. Patients with a history of recent alcohol or substance abuse (< 1 year)
21. Patients with a history of non-compliance with other therapies
22. Patients who have any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To assess toxicity of Etanercept (Enbrel) in children with Fanconi Anemia (FA) and early marrow failure. | 24 months
To assess efficacy of Etanercept (Enbrel) in improving hematopoiesis (i.e. peripheral counts) in patients with FA. | 24 months

SECONDARY OUTCOMES:
Correlation of biological studies to measure the impact of Etanercept (Enbrel) on Tumor Necrosis Factor - alpha (TNF-alpha) production. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stella M. Davies, MBBSPhd MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States